CLINICAL TRIAL: NCT00271622
Title: Neurodevelopmental and Behavioral Phenotyping Screening Protocol
Brief Title: The Neurodevelopmental and Behavioral Phenotyping Screening Protocol
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060065; 06-M-0065
Record Dates: First submitted 2005-12-31; First posted 2006-01-02 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-10

CONDITIONS: Neurologic Disorders; Autism; Neurodegenerative Disease; Neurobehavioral Manifestation
Keywords: Developmental Delay; Pediatric; Pervasive Developmental Disorder; Early Development; Healthy Control Subjects; Autism Spectrum Disorders; Healthy Volunteer; HV
MeSH Terms: conditions — Nervous System Diseases; Autistic Disorder; Neurodegenerative Diseases; Neurobehavioral Manifestations; Learning Disabilities; Child Development Disorders, Pervasive; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy volunteers: healthy volunteers
- individuals at risk: individuals with risk for psychiatric disorders or neurodevelopmental disorders, such as autism spectrum disorders.

SUMMARY:
The purpose of this protocol is to allow for the careful evaluation of healthy volunteers and individuals with risk for psychiatric disorders or neurodevelopmental disorders, such as autism spectrum disorder for specific protocols at NIH....

DETAILED DESCRIPTION:
The purpose of this protocol is to allow for the careful evaluation of healthy volunteers and individuals with risk for psychiatric disorders or neurodevelopmental disorders, such as autism spectrum disorders. The evaluations may be used to determine if the participant meets criteria for participation in research protocols at the National Institute of Mental Health (NIMH) and other collaborative investigations. Since the entry criteria for these protocols vary, the screening evaluations will also vary. Behavioral evaluations will also be done through this protocol for individuals participating in IRB-approved protocols being conducted by collaborating scientists at NIH. The evaluations might include: a psychiatric interview; a diagnostic interview; developmental and/or cognitive testing; ratings of other psychiatric symptoms; neuropsychological testing; a medical history; a physical exam; blood; and a request for medical records. Parents of minors will be interviewed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must be at least 6 weeks of age.
* Subjects or their parents must be competent to comprehend the purpose of the screening process and to provide written informed consent. Parents/guardians will sign the consent form, and both minors and adults (depending on results of capacity assessment) will be asked to assent only if it is determined that they understand their role in the study.
* Subjects must be willing to undergo an evaluation which may include a psychiatric interview; and medical, neurological, and laboratory examinations (as appropriate, such as renal and liver function tests, serum electrolytes, urinalysis, blood levels of psychotropic drugs, and urine drug screen for the presence of psychoactive drugs and drugs of abuse, as determined on a subject-to-subject basis).

EXCLUSION CRITERIA:

-Lack of appropriate consent: For minor patients, consent must be obtained from all legal guardians/caretakers, including both parents in separated or divorced families where there is shared legal custody of the child. In such cases, both parents must consent to the child s participation in this protocol.

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of healthy volunteers and individuals with risk for psychiatric disorders or neurodevelopmental disorders, such as autism spectrum disorders.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-02-27 (Actual)

PRIMARY OUTCOMES:
Screening evaluations such as a psychiatric interview; a diagnostic interview; developmental and/or cognitive testing; ratings of other psychiatric symptoms | Ongoing
  Screening evaluations such as a psychiatric interview; a diagnostic interview; developmental and/or cognitive testing; ratings of other psychiatric symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Genalynne C Mooneyham, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Farmer C, Adedipe D, Bal VH, Chlebowski C, Thurm A. Concordance of the Vineland Adaptive Behavior Scales, second and third editions. J Intellect Disabil Res. 2020 Jan;64(1):18-26. doi: 10.1111/jir.12691. Epub 2019 Oct 28. PMID 31657503
- [Derived] Manwaring SS, Mead DL, Swineford L, Thurm A. Modelling gesture use and early language development in autism spectrum disorder. Int J Lang Commun Disord. 2017 Sep;52(5):637-651. doi: 10.1111/1460-6984.12308. Epub 2017 Jan 24. PMID 28120370
- [Derived] Swineford LB, Guthrie W, Thurm A. Convergent and divergent validity of the Mullen Scales of Early Learning in young children with and without autism spectrum disorder. Psychol Assess. 2015 Dec;27(4):1364-78. doi: 10.1037/pas0000116. Epub 2015 Apr 20. PMID 25894712
- [Derived] Thurm A, Manwaring SS, Luckenbaugh DA, Lord C, Swedo SE. Patterns of skill attainment and loss in young children with autism. Dev Psychopathol. 2014 Feb;26(1):203-14. doi: 10.1017/S0954579413000874. Epub 2013 Nov 25. PMID 24274034
- [Derived] Joseph L, Thurm A, Farmer C, Shumway S. Repetitive behavior and restricted interests in young children with autism: comparisons with controls and stability over 2 years. Autism Res. 2013 Dec;6(6):584-95. doi: 10.1002/aur.1316. Epub 2013 Jul 18. PMID 23868881
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2006-M-0065.html